CLINICAL TRIAL: NCT05237154
Title: Secondary Effects of Intermittent Fasting and Physical Exercise on the Modulation of the Gut Microbiota, Body Composition and Inflammatory Process in Obesity.
Brief Title: Intermittent Fasting and Exercise: Effects on Gut Microbiota, Body Composition and Inflammation.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Sao Paulo (Other)
Collaborators: Fundação de Amparo à Pesquisa do Estado de São Paulo (Other Government); Coordenação de Aperfeiçoamento de Pessoal de Nível Superior. (Other Government)
Responsible Party: Principal Investigator, Ellen Cristini de Freitas, Principal Investigator, University of Sao Paulo
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Gut Microbiota-Obesity
Record Dates: First submitted 2022-01-20; First posted 2022-02-11 (Actual); Last update posted 2022-02-11 (Actual); Status verified 2022-02

CONDITIONS: Composition and Function of the Gut Microbiota Post Intervention; Metabolic and Inflammatory Variables Post Intervention
Keywords: Obesity; Gut microbiota; Intermittent fasting; High-intensity interval training; Metataxononic; Body composition
MeSH Terms: conditions — Obesity; Intermittent Fasting | interventions — Methods; High-Intensity Interval Training

STUDY DESIGN:
Intervention Model Description: Randomized clinical trial.
Masking Description: Participants will be randomly distributed into 3 groups: the intermittent fasting group (GIF) composed of individuals who will only perform the nutritional intervention for 8 weeks; the physical exercise group (GEX), composed of individuals who will perform only physical training for 8 weeks and the intermittent fasting group associated with physical exercise (GIF+EX), composed of individuals who will perform the nutritional intervention combined with physical training in the period of 8 weeks.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intermittent fasting (IF) (Experimental): Alternate-day intermittent fasting. Consumption of 25% of daily energy requirements on scheduled fasting days involving energy restriction for 2 non-consecutive days of the week and ad libitum feeding on the other 5 days of the week. Period: 8 weeks.
  Interventions: Other: Intervention with intermittent fasting.
- Exercise: High-Intensity Interval Training (HIIT) (Experimental): High intensity circuit training. Progressive training protocol 3x/week, for 8 weeks, with at least 1 day of rest between sessions and duration of 25 minutes each session - 4 minutes of initial warm-up, 18 minutes of the main part and 3 minutes of relaxation. First and second week: 30 second run and recovery time. Third and fourth week: 35-second runtime and 25-second recovery time. Fifth and Sixth Week: 40-second runtime and 20-second recovery time. Seventh and eighth weeks: 45-second runtime and 15-second recovery time.
  Interventions: Other: Intervention with high-intensity interval training.

INTERVENTIONS:
Other: Intervention with intermittent fasting. — Intervention with fasting protocol of alternate days 2 days a week and the other days with ad libitum consumption. Restricted food in 25% of the total daily needs on the days of the intermittent fasting protocol, with 18 hours of fasting and 6 hours of restricted feeding (18:6).
  Other Names: IF
  Arms: Intermittent fasting (IF)
Other: Intervention with high-intensity interval training. — Intervention with high-intensity interval training, 3x per week, with intensity maintained between 70-85% of maximum heart rate.
  Other Names: HIIT
  Arms: Exercise: High-Intensity Interval Training (HIIT)

SUMMARY:
Obesity and overweight affect around 2 billion people worldwide. Despite the growing prevalence, the treatment of obesity is still an obscure field and the impacts of this disease on the clinical and public health perspective are urgent. Studies have demonstrated a fundamental role of the gut microbiota in the pathogenesis of obesity and discuss the impacts of diet and physical exercise on the microbiome profile. However, the mechanisms involved in these processes, referring to strategies such as intermittent fasting associated with physical training, are still poorly explored and understood. It is believed that intermittent fasting combined with physical exercise can promote a remodeling of the composition and function of the microbiota and that the present investigation is promising in the prevention and treatment of obesity.

DETAILED DESCRIPTION:
Background: Obesity and overweight affect about 2 billion people worldwide. Despite the growing prevalence, the treatment of obesity is still an obscure field and the impacts of this disease on the clinical and public health perspective are urgent. Studies have demonstrated a fundamental role of the gut microbiota in the pathogenesis of obesity and discuss the impacts of diet and physical exercise on the microbiome profile. However, the mechanisms involved in these processes, referring to strategies such as intermittent fasting associated with physical training, are still poorly explored and understood. It is believed that intermittent fasting combined with physical exercise can promote a remodeling of the composition and function of the microbiota and that the present investigation is promising in the prevention and treatment of obesity. Methods: 60 obese women will participate in the study and will be randomly divided into 3 groups: 1) the intermittent fasting group, submitted to a diet for 8 weeks (n= 20); 2) the physical exercise group, submitted to physical training for 8 weeks (n= 20); and 3) intermittent fasting group associated with physical exercise, submitted to both interventions for 8 weeks (n= 20). All volunteers will perform collections and evaluations (pre and post intervention) of anthropometry, food consumption, indirect calorimetry to assess resting energy expenditure, body composition by BodPod®, blood collection for biochemical analysis and gene expression, collection of feces for the analysis of the intestinal microbiota and physical tests (Shuttle Walking Test, multiple repetition test and functional strength) for the exercise groups. Expected results: The synergistic effects of the proposed intervention are expected to improve gut microbiota and metabolic parameters in obese women.

ELIGIBILITY:
Inclusion criteria:

* Age between 18 and 40 years;
* Women;
* Have a regular menstrual cycle;
* Body weight below 120 kg;
* BMI between 30 kg/m2 and 40 kg/m2.

Exclusion Criteria:

* Individuals with any disease;
* Smokers;
* Alcoholics;
* Use regular medication;
* Medical impediment to the practice of physical activities;
* Carry out nutritional monitoring;
* Being in treatment for weight loss;
* Present some discomfort in long periods of fasting.

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2018-07-01 (Actual); Primary Completion 2018-12-15 (Actual); Study Completion 2019-01-30 (Actual)

PRIMARY OUTCOMES:
Anthropometric changes (Body weight) | eight weeks
  Changes in body weight (kilograms - Kg) pre and post intervention.
Anthropometric - height assessment (meters) | eight weeks
  Height measured in meters
Anthropometric changes (BMI) | eight weeks
  Changes in body mass index (evaluated through a calculation that combines weight measured in kilograms divided by height in meters squared - BMI in kg/m^2) evaluated pre and post intervention.
Anthropometric changes (Circumferences) | eight weeks
  Changes in waist, abdominal, and hip circumferences (centimeters) evaluated pre and post intervention.
Body composition changes | eight weeks
  Changes in fat-free mass and fat mass evaluated pre and post intervention by whole-body air displacement plethysmography method, BodPod® .
Dietary intake changes | eight weeks
  Completion of the food record of three non-consecutive days, one day of the week that included the intermittent fasting protocol, another day of the week with ad libitum and a weekend day. This evaluation will take place pre-intervention, in the fourth week and after the intervention. Assessment of caloric intake, macronutrients and fiber evaluated pre and post intervention (Dietwin® software - São Paulo, Brazil).
Indirect calorimetry assessment | eight weeks
  Changes in resting metabolic rate (RMR) evaluated pre and post intervention by indirect calorimetry.
Indirect calorimetry assessment (energetic substrates) | eight weeks
  Changes in oxidation of substrates (lipids and carbohydrates) evaluated pre and post intervention by indirect calorimetry.
Changes in total cholesterol and lipid fractions | eight weeks
  Changes in total cholesterol, triglycerides, HDL-cholesterol and LDL-c evaluated pre and post intervention, quantified by Total Liquiform Cholesterol Kit, HDL Cholesterol Kit and Liquiform Triglycerides Kit, from Labtest diagnóstica®, using an enzymatic system and absorbance spectrophotometer.
Changes in plasma cytokines | eight weeks
  Changes in serum levels of cytokines IL-15, IL-10, TNF-α adiponectin, resistin, adipsin/Factor D, fetuin-A and C-reactive protein evaluated pre and post intervention, by MILLIPLEX® Kit.
Changes in nitrogen balance | eight weeks
  Determination of urinary nitrogen by chemiluminescence method. 24-hour urine analysis evaluated pre and post intervention. Calculation of nitrogen balance by a equation.
Changes in concentration of short-chain fatty acids (acetate, propionate, and butyrate) | eight weeks
  Quantification of short-chain fatty acids using stool samples, evaluated pre and post intervention, by gas chromatography method.
Changes in gut microbiota_Extraction and DNA sequencing and library preparation. | eight weeks
  Total fecal DNA extraction using the QIAamp 96 PowerFecal kit (Mobio-QIAGEN). Regions of interest V2-V3, V3-V4 and V4-V5 present in the extracted total DNA. Amplification and preparation of libraries according to the Illumina® kit protocol. 16S sequencing by Illumina® company's MiSeq platform. Metataxonomic analysis of 16S rDNA sequences by bioinformatics. Assessments analyzed pre and post intervention.
Changes in aerobic performance | eight weeks
  Physical tests performed pre and post intervention to assess aerobic physical fitness by incremental test adapted from Shuttle Walking.
Changes in strength performance | eight weeks
  Maximum dynamic muscular strength by test of multiple maximum repetitions (RM) in the leg press 45° and in the bench press.
Changes in strength performance | eight weeks
  Assessment of changes in maximal isometric muscle strength of the dorsal region and handgrip by dynamometry.
Changes in strength performance | eight weeks
  Strength endurance capacity by 1-minute functional tests (squat, free squat and push-up).

CONTACTS AND LOCATIONS:
Locations (2):
- Brazil (2):
  - University of São Paulo, School of Physical Education and Sports of Ribeirão Preto., Ribeirão Preto, São Paulo
  - Gabriela Batitucci, Ribeirão Preto, São Paulo

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Batitucci G, Almeida OG, De Martinis ECP, Solar I, Cintra DE, de Freitas EC. Intermittent fasting and high-intensity interval training do not alter gut microbiota composition in adult women with obesity. Am J Physiol Endocrinol Metab. 2024 Sep 1;327(3):E241-E257. doi: 10.1152/ajpendo.00310.2023. Epub 2024 Jun 26. PMID 38922577
- [Derived] Batitucci G, Faria Junior EV, Nogueira JE, Brandao CFC, Abud GF, Ortiz GU, Marchini JS, Freitas EC. Impact of Intermittent Fasting Combined With High-Intensity Interval Training on Body Composition, Metabolic Biomarkers, and Physical Fitness in Women With Obesity. Front Nutr. 2022 May 26;9:884305. doi: 10.3389/fnut.2022.884305. eCollection 2022. PMID 35694163